CLINICAL TRIAL: NCT03967743
Title: Application of a Systematic Developmental Assessment to a Novel Population: Infants With Rare Genetic Disorders
Status: Recruiting | Type: Observational
Sponsor: Boston Children's Hospital (Other)
Responsible Party: Principal Investigator, Monica Wojcik, Instructor in Pediatrics, Boston Children's Hospital
Other Study IDs: IRB-P00031382
Record Dates: First submitted 2019-05-28; First posted 2019-05-30 (Actual); Last update posted 2024-06-21 (Actual); Status verified 2024-06

CONDITIONS: Genetic Disease; Genetic Syndrome; Genetic Predisposition to Disease; Development, Infant; Development, Child
Keywords: Genetics; Infant Development
MeSH Terms: conditions — Genetic Diseases, Inborn; Genetic Predisposition to Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Infants with rare genetic disorders: This is a prospective, registry study of infants with genetic disorders being seen clinically in the NICU GraDS program.

SUMMARY:
The main objective of this study is to apply a well-established model of developmental surveillance (which evolved to characterize the outcomes of very low birth weight infants) to infants with genetic disorders. A novel clinical model for infants with rare genetic disorders has been created as a joint initiative between the Division of Newborn Medicine's NICU Growth and Developmental Support Programs (NICU GraDS) program and the Division of Genetics at Boston Children's Hospital (BCH). This study plans to enroll patients with genetic syndromes seen in this clinic into a prospective, longitudinal study in order to characterize their developmental profiles and needs.

DETAILED DESCRIPTION:
The main objective of this study is to apply a well-established model of developmental surveillance (which evolved to characterize the outcomes of very low birth weight infants) to infants with genetic disorders. A novel clinical model for infants with rare genetic disorders has been created as a joint initiative between the Division of Newborn Medicine's NICU Growth and Developmental Support Programs (NICU GraDS) program and the Division of Genetics at Boston Children's Hospital (BCH). This study plans to enroll patients with genetic syndromes seen in this clinic into a prospective, longitudinal study in order to characterize their developmental profiles and needs. Related factors such as quality of life and parental stress will also be assessed which will complement the evaluation of the role of a "developmental home" for these high risk infants. It is also hypothesized that gaps in care - mismatches between services received and services indicated based upon the developmental evaluation - will be identified. The results of this study will be used to inform future research efforts utilizing targeted approaches to improve developmental outcomes.

For infants with rare genetic disorders, the aims are as follows:

Aim 1: Characterize physical and psychosocial development using standardized longitudinal assessments.

Aim 2: Identify developmental service needs, prescription, and utilization.

Aim 3: Assess parental stress and health-related quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Eligible patients are infants under 4 years of age with genetic disorders undergoing developmental surveillance in the NICU GraDS program.

Exclusion Criteria:

* Children 4 years of age or older will be excluded.

Max Age: 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: This is a prospective, registry study of infants under 4 years of age with genetic disorders being seen clinically in the NICU GraDS program.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2019-08-26 (Actual); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Registry of infants with rare genetic disorders | Up to 18 years
  Study subjects will be followed in the NICU GraDS program until approximately 3 years of age, though there will be prospective review of medical records until a maximum age of 18 years.

CONTACTS AND LOCATIONS:
Overall Officials: Monica Wojcik, MD, Principal Investigator — Boston Children's Hospital
Locations (1):
- Boston Children's Hospital, Boston, Massachusetts, United States